CLINICAL TRIAL: NCT05241184
Title: Deriving Cardiac Reference Ranges at 3.0Tesla in Healthy Volunteers
Acronym: DECADENT-HV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Glasgow (Other)
Collaborators: NHS Greater Glasgow and Clyde (Other)
Responsible Party: Principal Investigator, Kenneth Mangion, Clinical Lecturer in Cardiology, University of Glasgow
Other Study IDs: GN20CA408
Record Dates: First submitted 2022-02-04; First posted 2022-02-15 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Healthy Volunteers
Keywords: cardiovascular magnetic resonance imaging; adenosine stress; parametric mapping; reference ranges; strain; healthy volunteers
MeSH Terms: conditions — Sprains and Strains

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Multiparametric stress CMR protocol — Multiparametric stress CMR protocol

SUMMARY:
Current MRI society guidelines recommend that reference ranges for specific imaging techniques (T1, T2 mapping, perfusion) are acquired on the MRI scanner that clinical work and research studies are being carried out on. We propose to undertake 32 multi parametric stress cardiac MRI scans on healthy volunteers (50% female, 50% male) over the age of 18 years. These measurements are not yet available for the 3.0T Prisma scanner at the Institute of Clinical Excellence (ICE), Queen Elizabeth University Hospital (QEUH). These values are essential to identify what is abnormal for people living in the west of Scotland.

DETAILED DESCRIPTION:
Imaging societies recommend that each MRI scanner has a locally-derived reference range for tissue characteristics, notably the longitudinal (T1) and transverse (T2) myocardial relaxation times, measured in milliseconds [16].

T1 reference values vary according to the magnetic field strength of the MRI scanner. T1 and T2 times (ms) are expectedly higher at 3.0T compared to 1.5T, in line with results obtained when working with the Siemens VERIO scanner based at the BHF Glasgow Cardiovascular Research Centre [17]. T2 values for 3.0T are, generally, not so well described and are known to vary between different manufacturers and systems.

A consensus statement by Society for Cardiovascular Magnetic Resonance (SCMR) endorsed by the European Association for Cardiovascular Imaging (EACVI) states that "Reference ranges should be generated from data sets that were acquired, processed, and analyzed in the same way as the intended application, with the upper and lower range of normal defined by the mean plus and minus 2 standard deviations of the normal data, respectively."[16] Myocardial blood flow measurements for both stress and rest are also distinct for individual scanners, especially at 3.0T. In fact, a number of centres have derived site specific and magnet specific reference ranges from healthy volunteers including 1)Stockholm, Sweden, 1.5T Siemens Avanto, 3.4 ± 0.7 ml/min/g [18] 2) Barts (London, UK) 3.0T Siemens Prisma, 3.00 +/-0.76 ml/g/min (unpublished data) and 3) Leeds, UK: 3.0T Siemens Prisma 2.89 ± 0.56 ml/g/min [19], 1.5T Philips Intera, 4.50 ± 0.91 ml/min/g[20] and studies are ongoing in sites such as Oxford (https://www.ouh.nhs.uk/research/patients/trials/stress-mri.aspx) . As can be seen, there is a wide spread of values and local reference ranges are urgently required (defined as stress MBF <2 standard deviations from the mean in healthy volunteers). These measurements are not yet available for the 3.0T Prisma scanner at the Institute of Clinical Excellence (ICE), Queen Elizabeth University Hospital (QEUH). These values are essential to identify what is abnormal for people living in the west of Scotland.

ELIGIBILITY:
Inclusion Criteria:

* Age 18≥years
* Capacity to provide written informed consent
* Able to comply with study procedures
* eGFR >45ml/min
* Vaccination status against SARS CoV-19 is not an exclusion criterion.

Exclusion Criteria:

* Contra-indication to CMR e.g. severe claustrophobia, metallic foreign body.
* Contra-indication to intravenous adenosine, i.e. severe asthma; long QT syndrome; second- or third-degree AV block and sick sinus syndrome.
* Lack of informed consent.
* Women who are pregnant, breast-feeding or of child-bearing potential (WoCBP) without a negative pregnancy test
* History of cardiovascular illness.
* Previous COVID-19 illness

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers aged at least 18 years with no prior medical history (including cardiovascular health problems, medication or systemic illness including COVID-19) will be invited to participate by i) contacting eligible participants from the Clinical research imaging volunteer bank ii) placing advertisements in public buildings (e.g. hospital, university). Vaccination status for SARS Coronavirus-19 is not an exclusion criterion.
  The other exclusion criteria include standard contraindications to MRI (e.g. metallic implants and metallic foreign body) and known or suspected pregnancy.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2021-11-10 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Peak stress myocardial blood (mg/ml/min) | Through study completion, on average <2years.
  Peak stress myocardial blood with adenosine vasodilator stress
Myocardial perfusion reserve | Through study completion, on average <2years.
  Myocardial perfusion reserve with adenosine vasodilator stress
Global and septal T1 (MOLLI, shMOLLI) T2 | Through study completion, on average <2years.
  reference ranges
Global and regional Circumferential strain (GCS) | Through study completion, on average <2years.
  using Displacement Encoding with Stimulated Echoes (DENSE) MRI.
Global and regional Longitudinal strain (GLS) | Through study completion, on average <2years.
  using Displacement Encoding with Stimulated Echoes (DENSE) MRI.

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Elizabeth University Hospital, Glasgow, Lanarkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Data sharing will be on reasonable request to the CI